CLINICAL TRIAL: NCT05591937
Title: Screening and Treatment for Anxiety & Depression (S.T.A.N.D): Alacrity Center Signature Project on Triaging and Adapting to Level of Care
Brief Title: S.T.A.N.D. Alacrity Center Signature Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michelle Craske, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P50MH126337 (NIH)
Record Dates: First submitted 2022-08-29; First posted 2022-10-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Depression; Anxiety
Keywords: personalized care; cognitive behavioral therapy; depression; anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptom Severity Decision-Making (Active Comparator): Using current symptom severity level to guide triaging and adapting level of care.
  Interventions: Behavioral: Self-Guided Online Prevention; Behavioral: Coach-Guided Online Cognitive Behavioral Therapy; Behavioral: Clinician-Delivered Psychological and Psychiatric Care
- Data-Driven Decision-Making (Experimental): Using data-driven algorithm that considers social determinants of mental health, early life adversity/stress, predisposing, enabling and need influences upon health services use, and comprehensive mental health status to guide triaging and adapting level of care.
  Interventions: Behavioral: Self-Guided Online Prevention; Behavioral: Coach-Guided Online Cognitive Behavioral Therapy; Behavioral: Clinician-Delivered Psychological and Psychiatric Care

INTERVENTIONS:
Behavioral: Self-Guided Online Prevention — An online wellness program that contains self-guided online CBT prevention strategies with demonstrated efficacy for depression and anxiety in college samples. Participants can learn skills for coping with common stressful experiences and build resilience at their own pace.
Behavioral: Coach-Guided Online Cognitive Behavioral Therapy — An online digital therapy program that consists of online CBT modules supported by coaches through video chats. The modules are evidence-based and formatted into a unified approach for depression, anxiety and worry, panic, social anxiety, trauma and sleep dysregulation (developed as part of the University of California, Los Angeles (UCLA) Depression Grand Challenge). Lessons are designed to respond to participants' specific symptoms. Participants can access the system through any personal device (phone, tablet or computer) and speak to a certified student coach through remote video chat.
Behavioral: Clinician-Delivered Psychological and Psychiatric Care — Evidence-based clinician-delivered CBT modules. Participants are connected to a team of clinicians who will evaluate participants' specific symptoms and create an individualized and tailored treatment plan. Treatment will include weekly sessions delivered through telehealth, and if deemed appropriate, participants may also have medication appointments.

SUMMARY:
The purpose of this study is to evaluate clinical decision-making algorithms for (a) triaging to level of care and (b) adapting level of care in a low income, highly diverse sample of community college students at East Los Angeles College (ELAC).

The target enrollment is 200 participants per year, for five years (N=1000). Participants are between the ages of 18 and 40 years and will be randomized into either symptom severity decision-making (SSD) or data-driven decision-making (DDD). Participants in each condition will be triaged to one of three levels of care, including self-guided online prevention, coach-guided online cognitive behavioral therapy, and clinician-delivered care. After initial triaging, level of care will be adapted throughout the entire time of the study enrollment. Participants will complete computerized assessments and self-report questionnaires as part of the study. The total length of participation is 40 weeks.

DETAILED DESCRIPTION:
Community colleges provide a critical pathway for workforce development and socio-economic gain, but this opportunity is mitigated by unmet need for mental health services, particularly for depression and anxiety, and particularly for racial/ethnic minority students. A scalable and effective system of care that manages mental health needs in concert with social mental health determinants is sorely needed. The Alacrity Center aims to implement the STAND system of care, which screens and treats anxiety and depression, for a highly diverse community college population. STAND triages to various level of care, ranging from self-guided online prevention, to coach-guided online cognitive behavioral therapy (CBT), to clinician-delivered care. After initial triaging, STAND makes adaptations to level of care throughout the entire time of study enrollment (e.g., moved up to a higher level of care during acute treatment). These triaging and adaptation decisions currently are based on current symptom severity. Such decisions can be optimized by comprehensive data-driven algorithms that predict the need for a particular level of care and for adaptation to level of care throughout treatment, and especially algorithms that are suited to the needs of underserved community college students who face substantial life stressors.

The overarching aim of the Signature Project is to evaluate clinical decision-making algorithms for (a) triaging to level of care and (b) adapting level of care in a low income, highly diverse sample of community college students at East Los Angeles College (ELAC). The end goal is to improve the effectiveness of STAND and to advance the science of personalized mental health. To do this, we will compare the standard approach that relies solely upon symptom severity to a data-driven approach to decision making that uses multivariate predictive algorithms comprised of baseline static and time-varying features from four overlapping and mutually reinforcing theoretical constructs: (1) social determinants of mental health (employment, income, housing & food security, discrimination, social support, race/ethnicity, acculturation, immigration status, gender, sexual orientation); (2) early adversity and life stressors; (3) predisposing, enabling and need influences upon health services use; and (4) comprehensive mental health status (depression, anxiety and suicide severity, comorbidities, neurocognitive functioning, emotion dysregulation, regulatory strategy use, treatment history and preferences, social, occupational, home and academic functioning). The overarching design is to randomize ELAC students to either symptom severity decision-making (SSD) or data-driven decision-making (DDD), and evaluate whether DDD improves adherence to treatment, symptoms, and functioning. Other aims of this project are to (a) identify distal and proximal risk factors for suicide and self-harm and (b) examine effects of the decision-making condition (SSD, DDD) on suicidality and self-harm outcomes.

Participants will be enrolled through recruitment efforts at ELAC. The target enrollment is 200 participants per year over five years (n = 1000 total). Participants are current ELAC student between the ages of 18-40. Predictors and outcomes will be assessed at baseline and either weekly or every 8 weeks until week 40. Multivariate prediction models will be used for initial level of care triaging and later adaptations of level of care based on a comprehensive set of variables that have been shown to drive current mental health needs. Participants will complete computerized assessments and self-report questionnaires. The total length of participation is 40 weeks.

Embedded components:

Component 1 to evaluate interventions aimed at improving STAND uptake: In October 2025 an embedded randomized component was launched within this parent trial to evaluate approaches for improving initial uptake and engagement with STAND at ELAC. Participants consented to the parent trial are additionally randomized 1:1:1 to receive one of 3 engagement intervention conditions: either 1) fotonovela 2) peer-led engagement navigator 3) enrollment as usual. There is no separate consent process nor additional eligibility criteria for this embedded component. Only participants consented to the Signature project are enrolled in this additional component.

Component 2 to evaluate evaluate a technology-enhanced suicide prevention intervention (TE-SPI): In July 2025 the project launched an embedded RCT to evaluate a technology-enhanced suicide prevention intervention (TE-SPI) that includes treatment components with demonstrated benefits in prior research (safety planning, BRITE app, caring contacts to support safety plan use, hope, and reasons for living) and leverages mobile technology to deliver just-in-time adaptive interventions when intervention is most needed. Using Tier II and Tier III participants consented to the Signature Project, which include students for whom additional intervention for SU/SH risk is indicated, this work will use a rapid prototyping and testing model to develop and test an adaptation of the existing BRITE app plus safety planning for the primarily Latinx ELAC population. We are randomizing consented Tier II and Tier III assigned Signature Project participants to evaluate 1) TE-SPI with STAND usual risk management protocol (URM) compared to 2) STAND URM alone. We hypothesize that TE-SPI will a) lead to increased treatment engagement/contacts (i.e. app, STAND); b) demonstrate safety as indicated by low levels of self-harm related adverse events (e.g. hospitalizations, ED visits); c) be associated with fewer SU/SH events and greater improvement in suicidality, compared to URM; and d) that intervention engagement/dose received will lead to reduced SU/SH behavior.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in the East Los Angeles College
* Either uninsured or covered by California Medicaid
* Own or have private access to internet to complete the assessments and online prevention and therapy programs

Exclusion Criteria:

* Unable to fully comprehend the consent form, respond adequately to screening questions, or maintain focus or to sit still during assessment
* Diagnosed with disorders requiring more specialized care (e.g., psychotic disorder, severe eating disorder, severe substance use disorder, severe neurological disorder), or marked cognitive impairment
* Currently treated by psychiatrist or psychologist during timeframe that the treatment is offered through STAND and is unwilling to fully transfer care to STAND

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Longitudinal trajectory of treatment adherence | Up to 40 weeks
  Number of clinician sessions or coaching lessons attended or the number of online lessons completed; number of missed/cancelled sessions with clinicians or coaches; number of times logged on and total time spent online (1 item each). Measured longitudinally to capture trajectory over the course of the treatment.
Baseline symptom severity for mental health | Baseline
  Computerized Adaptive Test - Mental Health (CAT-MH). Symptoms of depression and anxiety are assessed using item response theory (IRT), where a subset of items are selected from a pool of approximately 1000 questions based on participant impairment level. Higher scores reflect greater symptom severity. Measured prior to beginning treatment to capture baseline value.
Longitudinal trajectory of symptom severity for mental health | Up to 40 weeks
  Computerized Adaptive Test - Mental Health (CAT-MH). Symptoms of depression and anxiety are assessed using item response theory (IRT), where a subset of items are selected from a pool of approximately 1000 questions based on participant impairment level. Higher scores reflect greater symptom severity. Measured longitudinally to capture trajectory over the course of the treatment.
Baseline social, occupational, and home functioning | Baseline
  Work and Social Adjustment Scale: functioning at work/school, home, social, and leisure activities (5 items, scored on a 0 to 8 scale). Higher scores reflect better adjustment. Measured prior to beginning treatment to capture baseline value.
Baseline academic functioning | Baseline
  Healthy Minds Survey: grade point average and perceived impact of mental health on academic functioning (1 item each, scored on a 1 to 4 scale). Higher scores reflect poorer academic functioning. Measured prior to beginning treatment to capture baseline value.
Longitudinal trajectory of social, occupational, and home functioning | Up to 40 weeks
  Work and Social Adjustment Scale: functioning at work/school, home, social, and leisure activities (5 items, scored on a 0 to 8 scale). Higher scores reflect better adjustment. Measured longitudinally to capture trajectory over the course of the treatment.
Longitudinal trajectory of academic functioning | Up to 40 weeks
  Healthy Minds Survey: grade point average and perceived impact of mental health on academic functioning (1 item each, scored on a 1 to 4 scale). Higher scores reflect poorer academic functioning. Measured longitudinally to capture trajectory over the course of the treatment.
Suicide and self-harm | Up to 40 weeks
  Number of attempts of suicide and non-suicidal self harm (11 items, scored with yes/no). Higher scores reflect higher overall self harm risk.

SECONDARY OUTCOMES:
Demographic background | Baseline
  Healthy Minds Survey: age, sex assigned at birth, gender identity, sexual orientation, race/ethnicity, citizenship/immigration status (1 item each).
Language | Baseline
  Healthy Minds Survey: language most commonly spoken with friends (1 item).
Acculturative Stress | Baseline
  Societal, Attitudinal, Familial and Environmental Acculturative Stress Scale: validated with Black, Latino and Asian American samples, particularly among college samples (6 items, scored on a 1 to 4 scale). Higher scores reflect greater acculturative stress.
Major discrimination experiences | Baseline
  Major Experiences of Discrimination-Abbreviated: discrimination due to racial, ethnic, socioeconomic, gender or other reasons (12 items, scored on a 1 to 4 scale). Higher scores reflect more discrimination experiences.
Longitudinal trajectory of daily discrimination experiences | Up to 40 weeks
  Everyday Discrimination-Short Form: daily experiences of discrimination (6 items, scored on a 1 to 6 scale). Higher scores reflect more discrimination experiences. Measured longitudinally to capture trajectory over the course of the treatment.
Longitudinal trajectory of employment status | Up to 40 weeks
  Healthy Minds Survey (1 item). Measured at baseline and longitudinally to capture value prior to beginning treatment and trajectory over the course of the treatment.
Longitudinal trajectory of housing/food security and financial stress | Up to 40 weeks
  Assessment of food, housing, and financial needs (4 items, scored with 1 = yes and 0 = no). Higher scores reflect higher stress level. Measured at baseline and longitudinally to capture value prior to beginning treatment and trajectory over the course of the treatment.
Longitudinal trajectory of social support | Up to 40 weeks
  Medical Outcomes Social Support Survey: perceived level of social support (4 items, scored on a 1 to 5 scale). Higher scores reflect higher support level. Measured at baseline and longitudinally to capture value prior to beginning treatment and trajectory over the course of the treatment.
Early adversity | Baseline
  Adverse Childhood Experiences Questionnaire: exposure to early life adversity and maltreatment (10 items, scored with 1 = yes and 0 = no). Higher scores reflect greater adversity.
Life stress exposure | Baseline
  Youth Partners in Care Life Events Scale: exposure to 15 negative stressful life events in the past 6 months (18 items, scored with 1 = yes and 0 = no). Higher scores reflect more stress exposure.
Longitudinal trajectory of perceived life stress | Up to 40 weeks
  Perceived Stress Scale: exposure to ongoing life stress (1 item, scored on a 0 to 3 scale). Higher scores reflect greater perceived stress. Measured longitudinally to capture trajectory over the course of the treatment.
Beliefs about mental health treatment and stigma | Baseline
  Healthy Minds Survey: attitudes towards mental health treatment and perceived and personal stigma about receiving mental health treatment (8 items, scored on a 1 to 6 scale); adapted from the Perceived Devaluation-Discrimination scale. Higher scores reflect more stigmatizing beliefs.
Insurance status | Baseline
  Healthy Minds Survey: insurance status (1 item).
Willingness to pay | Baseline
  Modified Willingness to Pay Scale: maximum yearly amount that one is willing to pay for mental health treatment (1 item).
Perceived need | Baseline
  Healthy Minds Survey: perceived need for mental health services (1 item, scored on a 1 to 6 scale). Higher scores reflect lower perceived need.
Longitudinal trajectory of sleep quality | Up to 40 weeks
  Insomnia Severity Index: level of sleep quality and severity of insomnia (7 items, scored on a 1 to 5 scale). Higher scores reflect greater insomnia severity. Measured at baseline and longitudinally to capture value prior to beginning treatment and trajectory over the course of the treatment.
Longitudinal trajectory of substance use | Up to 40 weeks
  Computerized Adaptive Test - Substance Use Inventory (CAT-SUD). Symptoms are assessed using item response theory (IRT), where a subset of items are selected from a pool of approximately 1000 questions based on participant impairment level. Higher scores reflect greater substance use severity. Measured at baseline and longitudinally to capture value prior to beginning treatment and trajectory over the course of the treatment.
Other mental conditions | Baseline
  Screening Assessment for Guiding Evaluation-Self Report (SAGE-SR): computerized self-report assessment of Diagnostic Statistical Manual-5 (DSM-5) diagnoses.
Other medical conditions | Baseline
  Healthy Minds Survey: physical health (1 item).
Emotion dysregulation | Baseline
  Difficulties in Emotion Regulation Scale-Short Form: self-report of emotion dysregulation or affective instability, a trait associated with many forms of psychopathology and personality disorders (16 items, scored on a 1 to 5 scale). Higher scores reflect greater emotion dysregulation.
Verbal ability | Baseline
  The Vocabulary Test: a measure of verbal ability that correlates with Scholastic Aptitude Test (SAT) verbal scores. Administered digitally through the TestMyBrain neurocognitive test battery, which has been shown to have adequate psychometric properties according to the National Institutes of Health report. Higher scores reflect greater functioning in this domain.
Abstract reasoning | Baseline
  The Matrix Reasoning Test: a measure of intelligence quotient (IQ) and abstract reasoning that correlates with the SAT math scores. Administered digitally through the TestMyBrain neurocognitive test battery, which has been shown to have adequate psychometric properties according to the National Institutes of Health report. Higher scores reflect greater functioning in this domain.
Cognitive response | Baseline
  The Choice Reaction Time Test: a measure of cognitive processing, response selection and inhibition aspects of cognitive control. Administered digitally through the TestMyBrain neurocognitive test battery, which has been shown to have adequate psychometric properties according to the National Institutes of Health report. Higher scores reflect greater functioning in this domain.
Selective attention | Baseline
  The Gradual Onset Continuous Performance Test: a measure of sustained attention and response inhibition. Administered digitally through the TestMyBrain neurocognitive test battery, which has been shown to have adequate psychometric properties according to the National Institutes of Health report. Higher scores reflect greater functioning in this domain.
Processing speed | Baseline
  Digit Symbol Matching Test: a measure of processing speed. Administered digitally through the TestMyBrain neurocognitive test battery, which has been shown to have adequate psychometric properties according to the National Institutes of Health report. Higher scores reflect greater functioning in this domain.
Visuospatial information processing | Baseline
  Multiple Object Tracking Test: a measure of visuospatial attention and visual working memory. Administered digitally through the TestMyBrain neurocognitive test battery, which has been shown to have adequate psychometric properties according to the National Institutes of Health report. Higher scores reflect greater functioning in this domain.
Socioemotional information processing | Baseline
  Multiracial Emotion Identification Test: a measure of emotion recognition and social perception. Administered digitally through the TestMyBrain neurocognitive test battery, which has been shown to have adequate psychometric properties according to the National Institutes of Health report. Higher scores reflect greater functioning in this domain.
Mental health treatment history | Baseline
  Healthy Minds Survey: prior therapy, medications, and helpfulness (4 items).
Mental health treatment preference | Baseline
  Preference Scale: preference for online vs. clinician-delivered therapy (1 item).
Longitudinal trajectory of regulatory strategy use | Up to 40 weeks
  Modified brief cognitive emotion regulation questionnaire: self-report of emotion regulatory strategy use (9 items, scored on a 1 to 5 scale). Higher scores reflect more frequent use of regulatory strategies. Measured at baseline and longitudinally to capture value prior to beginning treatment and trajectory over the course of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Craske, Ph.D, Principal Investigator — University of California, Los Angeles; Kate Taylor, Ph.D, Principal Investigator — University of California, Los Angeles
Locations (1):
- East Los Angeles College, Los Angeles, California, United States

REFERENCES:
- [Derived] Wen A, Wolitzky-Taylor K, Gibbons RD, Craske M. A randomized controlled trial on using predictive algorithm to adapt level of psychological care for community college students: STAND triaging and adapting to level of care study protocol. Trials. 2023 Aug 9;24(1):508. doi: 10.1186/s13063-023-07441-7. PMID 37553688

DOCUMENTS (1):
  • Study Protocol (2026-01-26): https://cdn.clinicaltrials.gov/large-docs/37/NCT05591937/Prot_001.pdf